CLINICAL TRIAL: NCT00161395
Title: Randomized Trial of Fertility Awareness and Time to Pregnancy in Couples of Normal Fertility
Brief Title: Study of Time to Pregnancy in Normal Fertility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Joseph Stanford, M.D., Principal Investigator, University of Utah
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: K23HD001479 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2005-09

CONDITIONS: Fertility; Pregnancy
Keywords: fertility; pregnancy
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Preconception advice.
  Interventions: Behavioral: Preconception advice
- 2 (Experimental): Instruction in the Creighton Model Fertility Care System.
  Interventions: Behavioral: Instruction in the Creighton Model Fertility Care System

INTERVENTIONS:
Behavioral: Instruction in the Creighton Model Fertility Care System — Instruction in the Creighton Model Fertility Care System.
  Other Names: Fertility awareness instruction.
  Arms: 2
Behavioral: Preconception advice — Preconception advice for diet and frequency of intercourse.
  Arms: 1

SUMMARY:
The purpose of this study is to determine how long it takes couples of normal fertility to get pregnant once they begin to try, and whether instruction in fertility awareness can decrease time to pregnancy in these couples.

DETAILED DESCRIPTION:
Research has established that there are relatively few days of the menstrual cycle that have a substantial probability of pregnancy from coitus, and that there are prospective biomarkers that allow a woman or couple to identify these "fertile" days. However, it remains unclear how this knowledge may improve a couple's chances of conceiving.

All couples participating in this study must have a history of previous pregnancy together and no history suggesting subfertility. Participants in this study will be randomly assigned to one of two groups. One group will receive instruction about identifying the days when a woman is mostly likely to get pregnant from intercourse, using the Creighton Model FertilityCare System, and the other group will receive instructions about the menstrual cycle, fertility, and preparing for pregnancy. Randomization is stratified by age.

All participants will keep a daily fertility chart and use a computerized device called the Fertility Monitor with urine dipsticks to monitor hormones of the menstrual cycle.

The primary outcome is time to pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* couple with prior pregnancy within the past 8 years

Exclusion Criteria:

* any history that suggests subfertility
* any history that suggests a medical contraindication for pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2003-01; Primary Completion 2006-08 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time to Pregnancy | Up to one year.

SECONDARY OUTCOMES:
Distribution of coitus within "fertile" days of menstrual cycle | Seven menstrual cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Stanford, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Dept. Family and Preventive Medicine, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Stanford JB, Smith KR, Varner MW. Impact of instruction in the Creighton model fertilitycare system on time to pregnancy in couples of proven fecundity: results of a randomised trial. Paediatr Perinat Epidemiol. 2014 Sep;28(5):391-9. doi: 10.1111/ppe.12141. PMID 25225008